CLINICAL TRIAL: NCT05001633
Title: A Pilot Study to Assess the Impact of Exposure to Popular Media Content on Patients Living With Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 135462
Record Dates: First submitted 2021-07-19; First posted 2021-08-12 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Obesity
Keywords: obesity; media content
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: 2-arm parallel group
Who Masked: Participant
Masking Description: Participants will not know what group they are allocated to until the intervention is delivered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): modified media content experience
  Interventions: Behavioral: modified media content paradigm
- Control (Active Comparator): media content experience
  Interventions: Behavioral: control

INTERVENTIONS:
Behavioral: modified media content paradigm — media content
  Arms: Intervention
Behavioral: control — media content experience
  Arms: Control

SUMMARY:
This study will explore the impact of exposure to popular media content on patients living with obesity. Findings from this study will provide new insights that will extend current understanding of exposure to media portrayal. This is a proof of principle pilot study that will evaluate the feasibility of recruitment, randomisation, assessment procedures and implementation of the intervention with the aim to facilitate the planning and the conduct of a full-scale randomised controlled trial.

DETAILED DESCRIPTION:
This study will explore the impact of exposure to popular media content on patients living with obesity. Findings from this study will provide new insights that will extend current understanding of exposure to media portrayal. This is a proof of principle pilot study that will evaluate the feasibility of recruitment, randomisation, assessment procedures and implementation of the intervention with the aim to facilitate the planning and the conduct of a full-scale randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Female adults aged 18-65 years.
2. Body Mass Index equal or greater than 30 kg/m2.
3. Weight stable at time of recruitment, defined as less than 5% variation in body weight over the preceding 3 months.
4. Proficient in written and spoken English.
5. Able to comply with study protocol.
6. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Type 1 and type 2 diabetes (in view of altered circulated gut hormone profiles and gustatory function).
2. Smoking (in view of the fact that smoking affects salivary cortisol).
3. Diagnosed with uncontrolled severe depression.
4. Diagnosed with uncontrolled psychiatric disorder.
5. Previous bariatric surgery.
6. Acute illness or chronic conditions that may impact HPA including Cushing syndrome.
7. Known or suspected history of HIV, Hepatitis B or C or other blood-borne diseases (in view of safety regulations regarding exposure to blood products).
8. Currently using glucocorticoids.
9. Pregnancy or lactation.
10. Elevated self-perceived stress as assessed by the Perceived Stress Scale.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Not based on self-representation of gender identity
Enrollment: 20 (Estimated)
Dates: Start 2021-07-09 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Cortisol levels | up to 4 hours
  To characterise the effect of a modified media content upon cortisol secretion in people living with obesity.

SECONDARY OUTCOMES:
heart rate | up to 4 hours
  To characterise the impact of a modified media content on heart rate
systolic and diastolic blood pressure | up to 4 hours
  To characterise the impact of a modified media content on blood pressure
blood glucose | up to 4 hours
  To characterise the impact of a modified media content on blood glucose
salivary hormones | up to 4 hours
  To characterise the impact of a modified media content on salivary hormones - what hormones will be analysed will depend on the availability of assays and will be decided later on at the end of the study
inflammatory cytokines | up to 4 hours
  To characterise the impact of a modified media content on inflammatory cytokines - what cytokines will be analysed will depend on the availability of assays and will be decided later on at the end of the study
dietary intake | up to 4 hours
  To characterise the impact of a modified media content on dietary intake through the use of an online recalling diary called Intake24
experience | up to 4 hours
  To evaluate participants' experience through semi-structure interviews

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Undecided